CLINICAL TRIAL: NCT06563115
Title: A Randomized, Double-Blinded, Placebo-Controlled, Single and Multiple Ascending Dose Study in Overweight/Obese Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of (PEG)-BHD1028
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of (PEG)-BHD1028
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EncuraGen, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ECN1028-101
Record Dates: First submitted 2024-07-26; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blinded, Placebo-Controlled, Single and Multiple Ascending Dose Study
Who Masked: Participant, Investigator
Masking Description: Double: participant, investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo_Single Ascending Dose (Placebo Comparator): Participants received a single SC dose of placebo on Day 1
  Interventions: Other: Placebo
- Experimental (PEG)-BHD1028_Single Ascending Dose (Experimental): Participants received a single escalated SC dose of (PEG)-BHD1028 on Day 1
  Interventions: Drug: (PEG)-BHD1028 Single Ascending Dose
- Placebo_Multiple Ascending Dose (Placebo Comparator): Participants received SC doses of placebo once a day for 28 days
  Interventions: Other: Placebo
- Experimental (PEG)-BHD1028_Multiple Ascending Dose (Experimental): Participants received SC doses of (PEG)-BHD1028 once a day for 28 days
  Interventions: Drug: (PEG)-BHD1028 Multiple Ascending Dose

INTERVENTIONS:
Drug: (PEG)-BHD1028 Single Ascending Dose — 4, 8, 16, 32, and 64 μg/Kg
  Other Names: adiponectin receptor agonist
  Arms: Experimental (PEG)-BHD1028_Single Ascending Dose
Drug: (PEG)-BHD1028 Multiple Ascending Dose — 8, 16, and 32 μg/Kg
  Other Names: adiponectin receptor agonist
  Arms: Experimental (PEG)-BHD1028_Multiple Ascending Dose
Other: Placebo — Diluent
  Arms: Placebo_Multiple Ascending Dose; Placebo_Single Ascending Dose

SUMMARY:
Adiponectin has been known to play critical roles in various physio-regulatory processes, and adiponectin deficiency may contribute to insulin resistance. (PEG)-BHD1028 was developed as an agonist of adiponectin receptors.

This first-in-human study evaluates the safety, tolerability, pharmacokinetics, and pharmacodynamics of (PEG)-BHD1028 in healthy overweight/obese subjects with insulin resistance.

DETAILED DESCRIPTION:
(PEG)-BHD1028 is a peptide agonist to adiponectin receptors, AdipoR1 and R2, designed based on the active site of the hormone and receptor binding configurations. Various scientific and clinical research revealed that adiponectin deficiency is positively associated with pathophysiological conditions, including insulin resistance and inflammation. Despite the beneficial effects of adiponectin, the hormone could not be developed into a therapeutic agent because of the complications in controlling post-transcriptional modifications.

This study investigates the safety and tolerability of (PEG)-BHD1028 after a single ascending dose (SAD) of a placebo, 4, 8, 16, 32, and 64 μg/Kg and multiple ascending doses (MAD) of a placebo, 8, 16, and 32 μg/Kg for 28 days following Q.D. injection subcutaneously in the healthy obese/overweight subjects. The pharmacokinetics (PK) and pharmacodynamics (PD) are also evaluated following single and multiple doses and multiple doses, respectively. The changes in the inflammatory biomarkers are explored during the 28 days as a part of the MAD portion study.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c < 6.5 % by local laboratory analysis (one retest is permitted)
* Body Mass Index (BMI) ≥ 27 kg/m2
* HOMA-IR ≥ 1.8
* Female subjects must be non-pregnant and non-lactating, and females of childbearing potential must have used a stable regimen of highly effective contraceptive methods (for at least 2 months prior to the Screening) that they were willing to continue for at least 30 days after the last dose of the study drug.
* Male subjects must be surgically sterile, abstinent or, if engaged in sexual relations with a woman of childbearing potential, the subject and his partner must use an acceptable method of contraception for at least 90 days after the last dose of the study drug.
* Ability and willingness to comply with all protocol procedures
* Ability to provide written informed consent

Exclusion Criteria:

* History of type 1 or 2 diabetes mellitus (T1DM, T2DM)
* Systolic blood pressure > 159 mm Hg or diastolic blood pressure > 99 mmHg at ----Screening (reading may be repeated on a different day)
* Treatment with antihypertensive medication or statins if the medication was not stable during the 2 months prior to Screening
* Treatment with thyroid hormones was not stable during the 3 months prior to Screening
* History of any weight control treatment, including over-the-counter and herbal medication and supplements, or any medication with a labeled indication for weight loss or weight gain within 30 days prior to Screening
* History of gastrointestinal surgery for obesity that may induce malabsorption, or any malabsorption disorder, or clinically significant (C.S.) ongoing gastrointestinal disorders (including gastroparesis, peptic ulcers, and severe gastrointestinal reflux disease)
* History of symptomatic heart failure (New York Heart Association class II, III, or IV), myocardial infarction, unstable angina, transient ischemic attack, cerebral infarct, cerebral hemorrhage, or invasive cardiovascular procedure (including coronary artery bypass grafting [CABG] and percutaneous coronary intervention [PCI]) within 6 months of Screening
* Presence of CS ECG findings (including corrected Q.T. interval using Fridericia's formula [QTcF] > 450 msec for males, QTcF > 470 msec for females, left bundle branch block [LBBB]) at Screening, or cardiac arrhythmia requiring medical or surgical treatment within 6 months prior to Screening
* Presence of any C.S. physical, laboratory, ECG finding, or medical condition (including moderate to severe osteoarthritis or other C.S. rheumatological disease), that (in the opinion of an Investigator) may interfere with any aspect of the study conduct or interpretation of results
* Estimated glomerular filtration rate [eGFR] < 60 mL/min/1.73 m2 at Screening (using the Modification of Diet in Renal Disease [MDRD] equation)
* Clinically significant disease (within the last five years) of the gastrointestinal, cardiovascular, hepatic, neurological, renal, pancreatic, immunological, dermatological, endocrine, genitourinary or hematological system
* Chronic liver disease, HIV, HBV- or active HCV infection, or a positive test at Screening
* History of mental handicap, major depression, suicidal behavior or attempts, or other psychiatric disorders requiring medical treatment (within 2 years of Screening), including selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), antipsychotics, lithium, or other psychiatric disorders including eating disorders and seizures
* Fasting triglycerides > 500 mg/dL or alanine aminotransferase (ALT) and/or (aspartate aminotransferase ) AST d> 2 x upper limit of normal (ULN) (a single retest of triglycerides, ALT, or AST was allowed)
* Use of any drugs that were known to interfere with glucose or insulin metabolism, including oral corticosteroids, glucagon-like peptide-1 (GLP-1) receptor agonists, monoamine oxidase (MAO) inhibitors, and growth hormone, or use of non-prescription drugs within 7 days of first dosing
* Administration of vaccines/immunizations within 14 days prior to the initiation of dosing
* Major surgery within 8 weeks prior to Screening
* History of, or suspected allergy or hypersensitivity to the investigational product (I.P.) components
* History of any active infection within 14 days prior to Screening
* Participation in any other clinical interventional study receiving active treatment within 30 days or 5 half-lives prior to Screening, whichever was longer
* History of alcohol or illicit drug abuse, including marijuana, or a positive drug test at Screening
* History of alcohol abuse within approximately 1 year, or average daily alcohol intake >2 drinks for men and > 1 drink of alcoholic beverages for women, or positive alcohol breath test at Screening
* Daily use of more than 15 cigarettes/week or equivalent use of any tobacco product within 6 weeks prior to Screening, or inability to abstain from smoking during the study
* Existence of any surgical or medical condition that, in the judgment of an Investigator, might interfere with the absorption, distribution, metabolism, or excretion of the IP
* A history of fainting from blood collections or vasovagal syncope
* Any anticipated procedures that might have interfered with compliance or completion of the study
* Donation or loss of > 500 mL of blood or blood product within 56 days prior to Screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-06-23 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of (PEG)-BHD1028 -Single ascending dose as measured by TEAEs | Baseline to Day 3
  Treatment emergent adverse events (including clinical AEs and Lab AEs) after a single dose of (PEG)-BHD1028 (including clinical AEs and Lab AEs) of (PEG)-BHD1028
Safety and tolerability of (PEG)-BHD1028 -Multiple ascending dose as measured by TEAEs | Baseline to Day 29
  Treatment emergent adverse events (including clinical AEs and Lab AEs) after multiple doses of (PEG)-BHD1028

SECONDARY OUTCOMES:
Pharmacokinetics of (PEG)-BHD1028 after a single dose, Cmax | pre-dose, and at 30 min, 1 hr, 2 hr, 4 hr, 8 hr, 12 hr, and 24 hr after the single dose
  Maximum plasma concentration of (PEG)-BHD1028
Pharmacokinetics of (PEG)-BHD1028 after a single dose, Tmax | pre-dose, and at 30 min, 1 hr, 2 hr, 4 hr, 8 hr, 12 hr, and 24 hr after the single dose
  Time to reach Maximum plasma concentration of (PEG)-BHD1028
Pharmacokinetics of (PEG)-BHD1028 after a single dose, t1/2 | pre-dose, and at 30 min, 1 hr, 2 hr, 4 hr, 8 hr, 12 hr, and 24 hr after the single dose
  Time to reach apparent (PEG)-BHD1028 apparent terminal half life
Pharmacokinetics of (PEG)-BHD1028 after a single dose, AUClast | pre-dose, and at 30 min, 1 hr, 2 hr, 4 hr, 8 hr, 12 hr, and 24 hr after the single dose
  Area under the (PEG)-BHD1028 concentration -time curve up to the last measurable concentration in serum
Pharmacokinetics of (PEG)-BHD1028 after a single dose, AUCinf | pre-dose, and at 30 min, 1 hr, 2 hr, 4 hr, 8 hr, 12 hr, and 24 hr after the single dose
  AUCinf Area under the (PEG)-BHD1028 concentration -time curve up extrapolated to infinity
Pharmacokinetics of (PEG)-BHD1028 after a single dose, CL/F | pre-dose, and at 30 min, 1 hr, 2 hr, 4 hr, 8 hr, 12 hr, and 24 hr after the single dose
  CL/F Apparent clearance of the drug calculated as dose of drug divided by the AUC
Pharmacokinetics of (PEG)-BHD1028 after a single dose, Vd/F | pre-dose, and at 30 min, 1 hr, 2 hr, 4 hr, 8 hr, 12 hr, and 24 hr after the single dose
  Apparent Volume of distribution calculated as Total administered dose/initial plasma concentration
Pharmacokinetics of (PEG)-BHD1028 after multiple doses, Cmax | pre-dose, and post dose on Day 1, Day 14 and Day 28
  Maximum plasma concentration of (PEG)-BHD1028
Pharmacokinetics of (PEG)-BHD1028 after multiple doses, Tmax | pre-dose, and post dose on Day 1, Day 14 and Day 28
  Time to reach Maximum plasma concentration of (PEG)-BHD1028
Pharmacokinetics of (PEG)-BHD1028 after multiple doses, Cav,ss | pre-dose, and post dose on Day 1, Day 14 and Day 28
  Average plasma concentrate at steady state
Pharmacokinetics of (PEG)-BHD1028 after multiple doses, AUCtau | pre-dose, and post dose on Day 1, Day 14 and Day 28
  Area under the (PEG)-BHD1028 concentration -time curve up to the last dose
Pharmacokinetics of (PEG)-BHD1028 after multiple doses, t1/2 | pre-dose, and post dose on Day 1, Day 14 and Day 28
  Time to reach (PEG)-BHD1028 apparent terminal half life
Pharmacokinetics of (PEG)-BHD1028 after multiple doses, CLss/F | pre-dose, and post dose on Day 1, Day 14 and Day 28
  Apparent plasma clearance of drug after extravascular administration at steady state
Pharmacokinetics of (PEG)-BHD1028 after multiple doses, Vd/F | pre-dose, and post dose on Day 1, Day 14 and Day 28
  Apparent volume of distribution after extravascular administration
Pharmacokinetics of (PEG)-BHD1028 after multiple doses, Rac(Cmax) | post dose on Day 1 and Day 28
  Accumulation ratio calculated as Cmax (day 28)/ Cmax (day 1)
Pharmacokinetics of (PEG)-BHD1028 after multiple doses, Rac(AUC) | post dose on Day 1 and Day 28
  Accumulation ratio calculated as AUC0-t (day 28)/ AUC0-t (day 1)
Pharmacodynamics of (PEG)-BHD 1028 after multiple doses as measured by Insulin C -peptide | Day -1 and Day 28
  Insulin c-peptide as assessed by the net AUC at baseline and the percentage change from baseline. Responders defined as subjects which exhibited a reduction in insulin c-peptide AUC during the Mixed Meal Tolerance Test (MMTT) of at least 15% from Day -1 to Day 28.
Pharmacodynamics of (PEG)-BHD 1028 after multiple doses as measured by insulin | Day -1 and Day 28
  Insulin AUC as assessed by the net AUC at baseline and the percentage change from baseline during the Mixed Meal Tolerance Test (MMTT).
Pharmacodynamics of (PEG)-BHD 1028 after multiple doses as measured by glucose | Day -1 and Day 28
  Fasting plasma glucose (FPG), Post-prandial glucose (PPG), and glucose AUC assessed during the Mixed Meal Tolerance Test (MMTT).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Kankam, MD, Principal Investigator — Altasciences Clinical
Locations (1):
- Altasciences Clinical, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No